CLINICAL TRIAL: NCT04602065
Title: Evaluation of Safety and Efficacy of IBI318 Monotherapy for Relapsed/Refractory Extranodal NK/T Cell Lymphoma (Nasal Type), a Multicenter, Open-label Phase Ib/II Trial
Brief Title: Evaluation of Safety and Efficacy of IBI318 Monotherapy for Relapsed/Refractory Extranodal NK/T Cell Lymphoma (Nasal Type) Trial
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to the company's development strategy adjustment, Innovent Biologics has decided not to continue this study after consultation with investigators.
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI318B201
Record Dates: First submitted 2020-09-30; First posted 2020-10-26 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Extranodal NK/T Cell Lymphoma, Nasal Type
Keywords: ENKTL
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Previously received anti-PD1/PD-L1 antibodies (Experimental): Patients previously received anti-PD1/PD-L1 antibodies, except for those were primarily refractory to them.
  Interventions: Drug: IBI318(Recombinant human anti-PD1/PD-L1 bispecific antibody)
- Patients previously never received anti-PD1/PD-L1 antibodies (Experimental): Patients previously never received anti-PD1/PD-L1 antibodies.
  Interventions: Drug: IBI318(Recombinant human anti-PD1/PD-L1 bispecific antibody)

INTERVENTIONS:
Drug: IBI318(Recombinant human anti-PD1/PD-L1 bispecific antibody) — IBI318, 300mg, Q2W, Intravenous influsion.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of IBI318 monotherapy for relapsed/refractory extranodal NK/T cell lymphoma (nasal type).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically diagnosed as extra-nodal NK/T cell lymphoma (nasal type) according to WHO 2016 criteria;
2. Refractory and relapsed ENKTL patients, being relapsed is defined as re-occurrence of the same lymphoma lesions at the primary site or new sites after complete response (CR); being refractory is defined as having any of the following conditions: evaluated as stable disease (SD) or progression disease (PD) after 2 cycles of treatment; not being able to achieve partial response (PR) after 4 cycles of treatment; not being able to achieve complete response (CR) after 6 cycles of treatment. Patients that did not achieve remission, or relapsed/progressed after autologous stem cell transplantation (ASCT) could also be enrolled.
3. Patients must have received asparaginase-based chemotherapy previously (patients with phase I/II disease must have received radiotherapy previously).
4. With measurable foci, defined as: lymph nodes with long diameters>15mm，extra-nodal foci>10mm on CT scan;
5. ECOG PS (Eastern Cooperative Oncology Group Performance Status) point 0 or 1;

Exclusion Criteria:

1. Invasive NK cell leukemia;
2. Primary CNS lymphoma or CNS-involved lymphoma;
3. Patients with hemophagocytic syndrome;
4. Patients with lymphoma invading large pulmonary vessels;
5. Patients primarily resistant to anti-PD1,PD-L1,PD-L2 antibodies (generally considered as those received anti- PD1,PD-L1,PD-L2 antibodies as monotherapy or in combination with chemotherapy, but did not achieve PR or CR in non-maintenance treatment).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
ORR(evaluated by the independent review committee according to Lyric 2016 criteria.) | After the last subject completed follow-up visit of up to 24 weeks
  To evaluate the objective response rate (ORR) of IBI318 monotherapy for relapsed/refractory extranodal NK/T cell lymphoma (nasal type).

SECONDARY OUTCOMES:
ORR | After the last subject completed follow-up visit of up to 24 weeks
  To evaluate the objective response rate (ORR) of IBI318 monotherapy for relapsed/refractory extranodal NK/T cell lymphoma (nasal type) determined by the investigators according to Lugano 2014 criteria and Lyric 2016 criteria
CR/PR | After the last subject completed follow-up visit of up to 24 weeks
  To evaluate the complete response (CR) rate and partial response (PR) rate of IBI318 monotherapy for relapsed/refractory extranodal NK/T cell lymphoma (nasal type)
DCR | After the last subject completed follow-up visit of up to 24 weeks
  To evaluate the disease control rate (DCR) of IBI318 monotherapy for relapsed/refractory extranodal NK/T cell lymphoma (nasal type)
TTR2016 criteria.) | After the last subject completed follow-up visit of up to 24 weeks
  To evaluate the time to response (TTR) of IBI318 monotherapy for relapsed/refractory extranodal NK/T cell lymphoma (nasal type)
DOR | After the last subject completed follow-up visit of up to 24 weeks
  To evaluate the duration of response (DOR) of IBI318 monotherapy for relapsed/refractory extranodal NK/T cell lymphoma (nasal type)
PFS | After the last subject completed follow-up visit of up to 24 weeks
  To evaluate the progression-free survival (PFS) and PFS rate at 12 months of IBI318 monotherapy for relapsed/refractory extranodal NK/T cell lymphoma (nasal type)
OS(evaluated by the investigators according to Lugano 2014 criteria and Lyric 2016 criteria.) | After the last subject completed follow-up visit of up to 24 weeks
  To evaluate the overall survival (OS) and OS at 12 months of IBI318 monotherapy for relapsed/refractory extranodal NK/T cell lymphoma (nasal type)
adverse events | from enrollment until the last patient finishes OS follow-up, or finishes 24-month treatment and corresponding safety follow-up, whichever comes first.
  To evaluate the safety profile of IBI318 monotherapy for relapsed/refractory extranodal NK/T cell lymphoma (nasal type)

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangdong, China